CLINICAL TRIAL: NCT06093113
Title: Development and Evaluation of a Mobile App to Provide Bereavement Support for Adolescents in Grief
Brief Title: Alba - a Mobile App to Provide Bereavement Support for Adolescents in Grief
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-04309-01
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Complicated Grief Disorder

STUDY DESIGN:
Intervention Model Description: Intervention group and active control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants will complete a web based pre-assessment and then be given access to the app "Alba" for two months followed by a web based post-assessment including questions regarding their experiences of using the app, and follow-up questionnaires.
  Interventions: Behavioral: Alba - Youth in grief
- Control group (Active Comparator): Participants will get access to a website containing information about grief and grief reactions.
  Interventions: Behavioral: Control website

INTERVENTIONS:
Behavioral: Alba - Youth in grief — The app will build on principles of cognitive behavioural theory and therapy (CBT) and contains five main sections: Learning, Self-assessment, Manage symptoms, Find support and a Personal space.
  Arms: Intervention group
Behavioral: Control website — The website will contain information about grief and grief reactions similar to some of the information given in the app.
  Arms: Control group

SUMMARY:
The goal of this two-armed randomised controlled trial is to evaluate a psychosocial self-management mobile app providing bereavement support to adolescents in grief. The main questions it aims to answer are:

1. How do adolescents in grief interact with and use the app?
2. How do bereaved adolescents perceive the usability of the app?
3. Is the intervention feasible?
4. How is the meaningfulness of using the app perceived among adolescents in grief and what effect do the adolescents perceive it to have on their grieving process and everyday life?
5. Does access to the app affect symptoms of grief, complicated grief, post-traumatic stress and depression among bereaved adolescents?

Participants will:

* Test the app (intervention group) or a website containing (control group) psychoeducation for 2 months
* Fill out online questionnaires regarding their mental health (baseline, post, 6 months, 12 months).
* Fill out an online questionnaire regarding the acceptability and usability of the app (intervention group)
* Be asked to participate in narrative interviews (intervention group)

Researchers will compare the intervention group with the control group to see if the app has an effect on bereaved adolescents mental health.

DETAILED DESCRIPTION:
The need for professional support is evident in teenagers' grief and approximately half of the bereaved teenagers in Sweden report feeling in need of some type of help or support. Some teenagers in bereavement find it hard to seek help or that seeking help is embarrassing. It could also be hard to recognise if and when they need help, as they might have a low level of knowledge regarding symptoms of grief. Children and teenagers in need of preventive interventions often do not receive the care they need, but effective preventive interventions can support bereaved teenagers to work through their grief adaptively and thus decrease the risk of the negative consequences and complications of loss, such as experiencing complicated grief, depression or post-traumatic stress. This may in turn reduce the need for clinical interventions for psychopathology.

A mobile app could be used as a platform for bereavement support and be a comforting aid available to bereaved teenagers without drawing the attention or knowledge of their peers. Web-based support can lead to younger people seek help at an earlier stage, due to lower stigmatisation. Mobile apps offer additional advantage over face-to-face and web-based interventions because of their availability, accessibility, the immediate support they can provide, and their anonymity (e.g., reducing barriers to seeking help for grief), low costs, and possible tailoring to the user (e.g., the user is in control over when and how to use the app). Therefore, mobile health (mHealth) offers a particularly great and ubiquitous platform for delivering mental health and supportive interventions to teenagers. However, there are few apps for children and teenagers and the benefit of mHealth for children is largely not evaluated. With this background, the research group has using Patient- and Public Involvement worked with 6 bereaved teenagers to develop a psychosocial self-management mobil app for adolescents in grief.

The overall purpose of this project is to evaluate a psychosocial self-management mobile app to provide bereavement support and self-help strategies to adolescents who have lost a parent or a sibling in fatal causes, in a randomised controlled trial. In order to evaluate the acceptability and feasibility of the intervention in bereaved teenagers, the trial will include a pilot phase during which results for recruitment, drop-out randomisation, retention rates and data collection will be used to identify and analyse potential issues with the trial before progression. Data related to the feasibility of the intervention and the accessibility of the app will in addition be collected during the post-assessment and be used to identify needed modifications for the app and the intervention. This data will, along with user-data, be used for evaluation of how bereaved adolescents use and engage with the app. To evaluate the effects of the app on bereaved adolescents mental health symptoms of grief, complicated grief, depression and post-traumatic stress will be measure at baseline, post 2 months of app/website usage, and at 6- and 12 months post randomisation, and compared between the intervention- and control group. Finally, to evaluate the meaningfulness of using the app and the self-perceived effect of the app intervention on bereaved adolescents' grieving process and everyday life, 10-15 participants of the intervention group will be asked to participate in narrative interviews. participants will be recruited using advertisement and in cooperation with non-profit organisations.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-19 years old
* Lost a parent or sibling to any cause of death at least one months ago
* Comprehend the Swedish language
* Have access to a mobile/smartphone

Exclusion Criteria:

* Loss occurred less than one month ago

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change (from baseline) in Traumatic Grief Inventory-Kids-Self report | 2, 6 and 12 months
  16-item, self-rated measure of complicated grief, total score ranges from 16 to 80, where higher score indicates more symptoms

SECONDARY OUTCOMES:
Change (from baseline) in Hogan Inventory for Bereavement- Short Form for Children and Adolescents | 2, 6 and 12 months
  21-item, self-rated measure of grief and personal growth, total score ranges from 10 to 50 for the subscale grief with a higher score indicating more symptoms, and a total score of 11 to 55 for the subscale personal growth.
Change (from baseline) in Child PTSD Symptom Scale | 2, 6 and 12 months
  27 item, self-rated measure of post-traumatic stress, total score ranges from 0 to 80 for the 20 symptom items, where a higher score indicating more symptoms
Change (from baseline) in Patient Health Questionnaire-9 | 2, 6 and 12 months
  9 item, self-rated measure of depression, total score ranges from 0 to 27, and a higher score indicates more symptoms

OTHER OUTCOMES:
Feasibility of the intervention and the application | 2 months
  Self-report questionnaire to assess feasibility.
Acceptability of the intervention and the application | 2 months
  Self-report questionnaire to assess user satisfaction and perceived helpfulness of the app.

CONTACTS AND LOCATIONS:
Overall Officials: Josefin Sveen, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code